CLINICAL TRIAL: NCT02849704
Title: Diagnosing Pancreatic-Based Malabsorption in Patients With Chronic Pancreatitis
Brief Title: Fat Malabsorption in Chronic Pancreatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: AbbVie (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Phoenix Indian Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-013001
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Chronic Pancreatitis
Keywords: Chronic Pancreatitis; Pancreatic Function; Reduced Exocrine Pancreatic Function; Pancreatic Insufficiency
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronic Pancreatitis (CP) Subjects (Experimental): CP subjects will fast for 12 hours prior to the malabsorption blood test (MBT) testing, consume the MBT breakfast meal following this fast, have blood drawn (MBT, vitamins A, D, E and K, zinc, selenium, and prealbumin) prior to MBT breakfast consumption and each hour for 8 hours after consumption, consume a low-fat study lunch, eat a moderate fat diet for 4 days during home diet and stool collection, maintain a 3-day food record, collect stool over 72 hours, have body size and composition assessment, complete quality of life questionnaires, home environment and health questionnaires, and adverse events diary.
  Subjects will take Creon36™ for 9 days.
  Subjects will have two study visits, one before and one after treatment initiation with Creon36™. Both visits will be identical with the exception of completion of questionnaires and fecal elastase assessment (only Visit 1).
  Interventions: Drug: Creon36™
- Healthy Controls (No Intervention): Healthy controls will fast for 12 hours prior to the malabsorption blood test (MBT) testing, consume the MBT breakfast meal following this fast, have blood drawn (MBT, vitamins A, D, E and K, zinc, selenium, and prealbumin) prior to MBT breakfast consumption and each hour for 8 hours after consumption, consume a low-fat study lunch, eat a moderate fat diet for 4 days during home diet and stool collection, maintain a 3-day food record, collect stool over 72 hours, have body size and composition assessment, complete quality of life questionnaires, home environment and health questionnaires, and adverse events diary. Controls will only have 1 study visit and receive no intervention.

INTERVENTIONS:
Drug: Creon36™ — Creon36™ delayed-release capsules, a pancreatic enzyme preparation, is an FDA approved medication. Subjects with chronic pancreatitis (CP) will take Creon36™ for nine days, at a daily dose of 72,000 lipase units per meal (two capsules) and 36,000 units per snack (one capsule), with each capsule containing 36,000 lipase units. Subjects will take Creon36™ for three days prior to Visit 2, the day of Visit 2 and then for five days after the visit until they have completed stool collections.
  Other Names: Pancrelipase; CREON
  Arms: Chronic Pancreatitis (CP) Subjects

SUMMARY:
The objective of this study is to evaluate the malabsorption blood test (MBT), stool coefficient of fat absorption (CFA) and stool bomb calorimetry (BC) methods as potential screening or diagnostic tests for reduced exocrine pancreatic function or pancreatic insufficiency (RPF/PI). A further objective is to determine the test responses before and after pancreatic enzyme medication administration (Creon36™) in the patients with chronic pancreatitis (CP).

DETAILED DESCRIPTION:
Reduced exocrine pancreatic function or pancreatic insufficiency (RPF/PI) contributes to poor clinical outcome in a number of diseases and conditions. The incidence, mechanism and substantial adverse clinical outcomes of pancreatic insufficiency (PI) are well known in patients with cystic fibrosis (CF), and the life sustaining role of pancreatic enzyme medication in CF care is well established. Much less is known about the incidence and impact of RPF/PI in patients with chronic pancreatitis (CP). Reliable non-invasive screening or diagnostic tests with acceptable patient burden are not available for RPF/PI.

This is a cohort study of subjects with CP who will be evaluated before and after pancreatic enzyme medication (Creon36™) administration. A cohort of healthy subjects will serve as a comparison group and will be evaluated only once.

Subjects with CP will receive Creon36™, a pancreatic enzyme medication, and fat and energy absorption will be evaluated using three methods: MBT, CFA, and BC before and after administration of Creon36™. Many patients with CP are at risk for RPF/PI yet they rarely undergo diagnostic testing. Pancreatic enzyme medication will likely improve clinical outcomes and quality of life in some of those with RPF/PI. A cohort of healthy volunteers will be evaluated with the three methods to provide essential comparison data to optimize the understanding and interpretation of the findings from the three methods and the RPF/PI cohort with CP. There will be no intervention for the healthy cohort.

ELIGIBILITY:
Inclusion Criteria (CP):

* Chronic pancreatitis diagnosis by gastroenterologist. Participants with CP will be characterized based on the TIGAR-O (toxic, genetic, autoimmune, recurrent, obstructive) etiology system, on pancreatic morphology (Cambridge criteria) when available, and on physiological state (exocrine and endocrine function) as recommended by the recent American Pancreatic Association Practice Guidelines4.
* Age 30-70 years old
* Evidence of at-risk for malabsorption including: 1) history of use of and response to pancreatic enzyme medication; 2) history of unintentional weight loss; 3) history of increased stools per week or fatty stools; and/or 4) other clinical signs or symptoms suggestive of fat malabsorption
* In usual state of health for past two weeks including no change in medications
* Able to consume a moderate fat diet for stool evaluations
* Able to participate in the study for about four weeks with two study visits

Inclusion Criteria (Healthy Volunteers):

* Age 30-70 years old
* No known chronic disease that would affect dietary intake or fat absorption
* In usual state of health for past two weeks, with stable medications, diet and weight
* BMI from 18-29
* Able to consume a moderate fat diet for stool evaluations
* Able to participate in the study for about one week with one study visit

Exclusion Criteria (CP):

* Evidence of normal fat absorption in medical record
* Medications that alter fat absorption (i.e. orlistat, other weight loss medications, ursodeoxycholic acid)
* Allergy to pork products
* History of intestinal blockage or fibrosing colonopathy
* History of gout, kidney disease, or high blood uric acid (hyperuricemia)
* Pregnancy or breast feeding

Exclusion Criteria (Healthy Volunteers):

* Evidence of fat malabsorption
* Medications that alter fat absorption (i.e. orlistat, other weight loss medications, ursodeoxycholic acid)
* Pregnancy or breast feeding

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Babette Zemel, PhD, Principal Investigator — Children's Hospital of Philadelphia; Virginia Stallings, MD, Study Director — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from academic medical centers in the Philadelphia region between August 2016 and November 2017. For the CP cohort, subjects were diagnosed with CP by a gastroenterologist based on criteria as recommended by the American Pancreatic Association (APA) Practice Guidelines.
Pre-assignment Details: There were no events between enrollment and assignment in either group. All subjects enrolled were assigned to the appropriate arm.
Groups:
- Chronic Pancreatitis (CP) Subjects: CP subjects will fast for 12 hours prior to the malabsorption blood test (MBT) testing, consume the MBT breakfast meal following this fast, have blood drawn (MBT, vitamins A, D, E and K, zinc, selenium, and prealbumin) prior to MBT breakfast consumption and each hour for 8 hours after consumption, consume a low-fat study lunch, eat a moderate fat diet for 4 days during home diet and stool collection, maintain a 3-day food record, collect stool over 72 hours, have body size and composition assessment, complete quality of life questionnaires, home environment and health questionnaires, and adverse events diary. This visit will be repeated after initiation of Creon36™.
Period: Washout Period - CP Subj on PERT - 3days
Arm/Group | Chronic Pancreatitis (CP) Subjects | Healthy Controls
Started (Subjects with a diagnosis of CP and who were taking PERT participated in this Period) | 11 | 0
Completed | 11 | 0
Not Completed | 0 | 0
Period: Baseline Assessments - All Subj - 7 Days
Arm/Group | Chronic Pancreatitis (CP) Subjects | Healthy Controls
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: Assessment on PERT - CP Subj - 16 Days
Arm/Group | Chronic Pancreatitis (CP) Subjects | Healthy Controls
Started | 24 | 0
Completed | 21 | 0
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Unable to complete study procedures | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Pancreatitis (CP) Subjects | Healthy Controls | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two healthy subjects were found after completion of assessments to have chronic illnesses not initially disclosed upon enrollment. Since they did not meet original inclusion criteria, they were dropped from analysis.
  years
    number analyzed (Participants) | 24 | 22 | 46
    (all) | 50.7 (9.6) | 43.4 (10) | 47.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two healthy subjects were found after completion of assessments to have chronic illnesses not initially disclosed upon enrollment. Since they did not meet original inclusion criteria, they were dropped from analysis.
  Participants
    number analyzed (Participants) | 24 | 22 | 46
    Female | 11 | 15 | 26
    Male | 13 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two healthy subjects were found after completion of assessments to have chronic illnesses not initially disclosed upon enrollment. Since they did not meet original inclusion criteria, they were dropped from analysis.
  Participants
    number analyzed (Participants) | 24 | 22 | 46
    Hispanic or Latino | 1 | 1 | 2
    Not Hispanic or Latino | 23 | 21 | 44
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two healthy subjects were found after completion of assessments to have chronic illnesses not initially disclosed upon enrollment. Since they did not meet original inclusion criteria, they were dropped from analysis.
  Participants
    number analyzed (Participants) | 24 | 22 | 46
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 9 | 9 | 18
    White | 13 | 12 | 25
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index Population: Two healthy subjects were found after completion of assessments to have chronic illnesses not initially disclosed upon enrollment. Since they did not meet original inclusion criteria, they were dropped from analysis.
  kg/m^2
    number analyzed (Participants) | 24 | 22 | 46
    (all) | 23.9 (3.6) | 25.6 (4.4) | 24.7 (4.0)
Fecal Elastase [Mean (Standard Deviation); unit: ug/g stool] — Population: This measure was only baseline for the CP group.
  ug/g stool
    number analyzed (Participants) | 24 | 0 | 24
    (all) | 169 (172) |  | 169 (172)
Coefficient of Fat Absorption [Mean (Standard Deviation); unit: % of dietary fat absorbed] — Population: Two healthy subjects were found after completion of assessments to have chronic illnesses not initially disclosed upon enrollment. Since they did not meet original inclusion criteria, they were dropped from analysis.
  Four subjects with CP did not have adequate stool collection (n=2) or fat intake (n=2) for a valid CFA test.
  % of dietary fat absorbed
    number analyzed (Participants) | 20 | 22 | 42
    (all) | 90.9 (12.8) | 95.4 (9.3) | 93.2 (9.2)
Bomb Calorimetry [Mean (Standard Deviation); unit: cal/g stool] — Population: 2 healthy subjects were found after assessment to have chronic illnesses not initially disclosed; they were dropped from analysis. 3 subjects were excluded from analysis due to uncertainty in test result (high variability in test runs). 1 subject with CP was excluded due to uncertainty, 2 were excluded due to inadequate stool collection.
  cal/g stool
    number analyzed (Participants) | 21 | 19 | 40
    (all) | 5728 (717) | 5171 (393) | 5463 (635)
HA AUC [Mean (Standard Deviation); unit: mg*h/dL] — Area under the curve for heptadecanoic acid Population: Of the subjects with CP, one did not complete the study meal for a valid test, and one was a significant outlier. Of the healthy subjects, two were deemed not healthy as previously explained, and two did not complete the study meal for a valid test.
  mg*h/dL
    number analyzed (Participants) | 22 | 20 | 42
    (all) | 8.3 (4.3) | 17.7 (10.3) | 12.7 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Malabsorption Blood Test: Difference in Mean HA AUC Between Groups: Subjects With CP Compared to Healthy Subjects
Description: The fat absorption pattern in CP subjects will be compared with healthy controls. Mean HA AUC will be calculated for the CP subjects and the healthy controls and compared to determine whether there is a difference in the fat absorption between the two groups.
Time Frame: 8 hours
Population: Two subjects with CP were excluded; one did not complete the study meal for a valid test, and one was a significant outlier calling into question the validity of the test. Of the 24 healthy controls, two were excluded from the study due to undisclosed chronic disease, and two subjects did not complete the study meal for a valid test.
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Chronic Pancreatitis (CP) Subjects | Healthy Controls
Number analyzed (Participants) | 22 | 20
mg*h/dL | 8.3 (4.3) | 17.7 (10.3)
Statistical Analysis 1: Comparison: Chronic Pancreatitis (CP) Subjects vs Healthy Controls; Test type: Superiority; p < 0.001, t-test, 2 sided — a priori threshold for significance: <0.05

2. Primary Outcome: Coefficient of Fat Absorption: Difference in Mean % Dietary Fat Absorption Between Groups: Subjects With CP Compared to Healthy Subjects
Description: The fat absorption pattern in CP subjects will be compared with healthy controls. Mean coefficient of fat absorption (% dietary fat absorbed) will be calculated for the CP subjects and the healthy controls and compared to determine whether there is a difference in the fat absorption between the two groups.
Time Frame: 72 hours
Population: Four subjects with CP were excluded; two did not consume enough fat for a valid test, one subject did not have adequate stool for analysis, and one subject was excluded due to an error in the lab processing stool. Of the 24 healthy controls, two were excluded from the analysis due to undisclosed chronic disease.
Measure: Mean (Standard Deviation); unit: % of dietary fat intake
Groups:
- Chronic Pancreatitis (CP) Subjects: As part of the primary assessment, CP subjects will eat a moderate fat diet for 4 days during home diet and stool collection, maintain a 3-day food record, and collect stool over 72 hours.
- Healthy Controls: Healthy controls will eat a moderate fat diet for 4 days during home diet and stool collection, maintain a 3-day food record, and collect stool over 72 hours.
Arm/Group | Chronic Pancreatitis (CP) Subjects | Healthy Controls
Number analyzed (Participants) | 20 | 22
% of dietary fat intake | 90.9 (12.8) | 95.4 (9.3)
Statistical Analysis 1: Comparison: Chronic Pancreatitis (CP) Subjects; Test type: Superiority; p > 0.05, t-test, 2 sided — a priori threshold for statistical significance <0.05

3. Primary Outcome: Bomb Calorimetry: Difference in Mean Stool Energy Loss Between Groups: Subjects With CP Compared to Healthy Subjects
Description: The energy absorption pattern in CP subjects will be compared with healthy controls. Mean calories per gram of stool will be calculated for the CP subjects and the healthy controls and compared to determine whether there is a difference in the stool energy loss between the two groups.
Time Frame: 72 hours
Population: Three subjects with CP were excluded; two did not consume enough fat for a valid test, one subject did not have adequate stool for analysis. Of the 24 healthy controls, two were excluded from the analysis due to undisclosed chronic disease, one did not provide adequate stool for analysis, and two results failed internal the validation protocol.
Measure: Mean (Standard Deviation); unit: calories/gram of stool
Arm/Group | Chronic Pancreatitis (CP) Subjects | Healthy Controls
Number analyzed (Participants) | 21 | 19
calories/gram of stool | 5728 (717) | 5171 (393)
Statistical Analysis 1: Comparison: Chronic Pancreatitis (CP) Subjects vs Healthy Controls; Test type: Superiority; p < 0.01, t-test, 2 sided — a priori threshold for statistical significance <0.05

4. Secondary Outcome: Bomb Calorimetry: Difference in Mean Energy Loss Between Groups: Subjects With CP Before and After Creon36™
Description: The energy absorption pattern in CP subjects before and after treatment with Creon36™ will be compared. Calories per gram of stool will be calculated for the CP subjects before and after the medication and compared to determine whether there is a difference in the stool energy loss in the same subjects between the two time points.
Time Frame: 72 hours
Population: Two subjects were excluded from follow-up due to inadequate stool provision. Two subjects were excluded due to failing the internal validation protocol.
Measure: Mean (Standard Deviation); unit: calories/gram of stool
Groups:
- Chronic Pancreatitis (CP) Subjects: For Visit 1, CP subjects will eat a moderate fat diet for 4 days during home diet and stool collection, maintain a 3-day food record, and collect stool over 72 hours.
  Subjects will take Creon36™ for 9 days at a daily dose of 72,000 lipase units per meal (two capsules) and 36,000 units per snack (one capsule), with each capsule containing 36,000 lipase units. Subjects will take Creon36™ for three days prior to Visit 2 and the day of Visit 2.
  Visit 2 will repeat Visit 1 study procedures.
Arm/Group | Chronic Pancreatitis (CP) Subjects
Number analyzed (Participants) | 20
calories/gram of stool | 5702 (691)
Statistical Analysis 1: Comparison: Chronic Pancreatitis (CP) Subjects; Test type: Superiority; p > 0.05, t-test, 2 sided — a priori threshold for statistical significance <0.05

5. Secondary Outcome: Malabsorption Blood Test: Difference in Mean HA AUC Between Groups: Subjects With CP Before and After Creon36™
Description: The fat absorption pattern in CP subjects before and after treatment with Creon36™ will be compared. Mean HA AUC will be calculated for the CP subjects before and after the medication and compared to determine whether there is a difference in the fat absorption in the same subjects between the two time points.
Time Frame: 8 hours
Population: For this paired analysis, twenty subjects had valid tests at both time points. Two subjects were excluded from baseline; one did not complete the study meal for a valid test, and one was a significant outlier calling into question the validity of the test. Two subjects were excluded from follow-up, as they did not complete the study meal or test.
Measure: Mean (Standard Deviation); unit: mg*h/dL
Groups:
- Chronic Pancreatitis (CP) Subjects: For Visit 1, CP subjects will fast for 12 hours prior to the malabsorption blood test (MBT) testing, consume the MBT breakfast meal following this fast, have blood drawn prior to MBT breakfast consumption and each hour for 8 hours after consumption, and consume a low-fat study lunch at hour 6 during the test.
  Subjects will take Creon36™ for 9 days at a daily dose of 72,000 lipase units per meal (two capsules) and 36,000 units per snack (one capsule), with each capsule containing 36,000 lipase units. Subjects will take Creon36™ for three days prior to Visit 2 and the day of Visit 2.
  Visit 2 will repeat Visit 1 study procedures.
Arm/Group | Chronic Pancreatitis (CP) Subjects
Number analyzed (Participants) | 20
mg*h/dL | 9.4 (4.2)
Statistical Analysis 1: Comparison: Chronic Pancreatitis (CP) Subjects; Test type: Superiority; p < 0.05, t-test, 2 sided — a priori threshold for statistical significance <0.05

6. Secondary Outcome: Coefficient of Fat Absorption: Difference in Mean % Dietary Fat Absorption Between Groups: Subjects With CP Before and After Creon36™
Description: The fat absorption pattern in CP subjects before and after treatment with Creon36™ will be compared. The % of dietary fat absorbed will be calculated for the CP subjects before and after the medication and compared to determine whether there is a difference in the fat absorption in the same subjects between the two time points.
Time Frame: 72 hours
Population: Two subjects were excluded from baseline due to inadequate dietary fat intake for a valid test, and one was excluded for inadequate stool provision. Three subjects were excluded at follow up for inadequate dietary information and stool provision. One subject was excluded from follow up due to lab error.
Measure: Mean (Standard Deviation); unit: % of dietary fat intake
Arm/Group | Chronic Pancreatitis (CP) Subjects
Number analyzed (Participants) | 17
% of dietary fat intake | 93 (8.8)
Statistical Analysis 1: Comparison: Chronic Pancreatitis (CP) Subjects; Test type: Superiority; p > 0.05, t-test, 2 sided — a priori threshold for statistical significance <0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the time period during which study procedures were undertaken. For healthy subjects, this includes the 7 days surrounding the assessment visit. For subjects with CP, this includes the 7 days surrounding the baseline assessment visit and the 9 days during which the subjects took Creon surrounding the second assessment visit.
Description: Adverse events were collected by personal interview during the visit itself, and by phone call after the completion of study procedures.
Arm/Group | Chronic Pancreatitis (CP) Subjects | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 7/24 | 3/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Pancreatitis (CP) Subjects (N=24) | Healthy Controls (N=24)
Abdominal Pain/Discomfort (Gastrointestinal disorders) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT02849704/Prot_SAP_000.pdf